CLINICAL TRIAL: NCT01181427
Title: A Blinded, Randomized, Placebo-Controlled Study in Healthy and HCV Genotype 1-infected Adults, to Evaluate the Safety, Tolerability, Antiviral Activity, Pharmacokinetics (Including the Effect of Food) and Resistance Profile of Single and Multiple Doses of ABT-267
Brief Title: Study of ABT-267 in Both Healthy Volunteers and Hepatitis C Virus (HCV) Genotype 1 Infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-116
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Single Ascending Dose (SAD) (Placebo Comparator): Healthy volunteers, receiving single ascending doses of ABT-267 or placebo.
  Interventions: Drug: ABT-267; Drug: Placebo
- Multiple Ascending Dose (MAD) (Placebo Comparator): Healthy volunteers, receiving multiple ascending doses of ABT-267 or placebo, OR, multiple doses of ABT-267 + single dose of a Cytochrome P450 inhibitor or placebo + single dose of a Cytochrome P450 inhibitor.
  Interventions: Drug: ABT-267; Drug: Placebo; Drug: Cytochrome P450 inhibitor
- Food Effect (FE) (Active Comparator): Healthy volunteers, receiving ABT-267, multi-dose, food effect.
  Interventions: Drug: ABT-267
- Antiviral Activity (Placebo Comparator): HCV genotype 1-infected treatment naïve subjects receiving multiple ascending doses of ABT-267 or placebo monotherapy for 3 days.
  Interventions: Drug: ABT-267; Drug: Placebo
- Resistance Monitoring (No Intervention): HCV genotype 1-infected treatment naïve subjects, receiving at least one dose of ABT-267 or placebo in the "Antiviral Activity" arm, follow-up to monitor resistance developed to ABT-267, no treatment and only blood samples will be collected
  Interventions: Procedure: Blood Sample Collection

INTERVENTIONS:
Drug: ABT-267 — See arm description
  Arms: Antiviral Activity; Food Effect (FE); Multiple Ascending Dose (MAD); Single Ascending Dose (SAD)
Drug: Placebo — See arms description
  Arms: Antiviral Activity; Multiple Ascending Dose (MAD); Single Ascending Dose (SAD)
Procedure: Blood Sample Collection — See arm description
  Arms: Resistance Monitoring
Drug: Cytochrome P450 inhibitor — See arm description
  Arms: Multiple Ascending Dose (MAD)

SUMMARY:
Study of ABT-267 in both healthy volunteers and Hepatitis C virus (HCV) genotype 1 infected subjects.

ELIGIBILITY:
Inclusion Criteria

Main Selection Criteria for Healthy Volunteers:

* Subject has provided written consent.
* Subject is in general good health.
* Females must be post-menopausal for at least 2 years or surgically sterile.
* Females must not be pregnant or breast-feeding. If male, subject is surgically sterile or practicing specific forms of birth control.

Main Selection Criteria for HCV Genotype 1-infected Volunteers:

* Subject has provided written consent.
* Subject has chronic HCV genotype 1 infection at screening.
* Liver biopsy within 3 years with histology.
* Females must be post-menopausal for at least 2 years or surgically sterile.
* Females must not be pregnant or breast-feeding. If male, subject is surgically sterile or practicing specific forms of birth control.
* Subject is in general good health, as perceived by the investigator, other than HCV infection.

Main Selection Criteria for Volunteers in the Resistance Monitoring Portion of the Study:

* Subject has provided written consent, has received at least one dose of ABT-267 or placebo in the study, and is considered suitable by the investigator to participate.

Exclusion Criteria

Main Exclusion Criteria for Healthy Volunteers:

* Positive test for HAV IgM, HBsAg, HCV Ab or HIV Ab.
* Clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder.
* Use of tobacco or nicotine-containing products with the 6-month period prior to study drug administration.
* Abnormal screening laboratory results.
* Significant sensitivity to any drug.
* Requirement for any over the counter and/or prescription medication, vitamins and/or herbal supplements on a regular basis.

Main Exclusion Criteria for HCV Genotype 1-infected Volunteers:

* Significant sensitivity to any drug.
* Positive HBsAg, HAV-IgM, and HIV Ab. Use of CYP enzyme inducers or inhibitors within 1 month of dosing.
* Clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid disease (except hypothyroidism on stable thyroid replacement therapy), or any uncontrolled medical illness or psychiatric disorder.
* Use of any medications (prescription and over-the counter) within 2 weeks prior to study drug dosing without prior approval by the Abbott Medical Monitor.
* Use of any vitamins or herbal supplements within 2 weeks prior to study drug dosing.
* Prior treatment with any investigational or commercially available anti-HCV agents.
* Abnormal screening laboratory results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Analysis of pharmacokinetic variables and mean change in HCV RNA level from baseline. | Up to 15 days or less
Analysis of safety measures including but not limited to tabulation of adverse events, physical exam, vital signs, ECGs, continuous cardiac monitoring, and clinical lab results (including chemistry, hematology and urine). | Update to 20 days or less

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Campbell, MD, Study Director — Abbott
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 42708, Orlando, Florida
  - Site Reference ID/Investigator# 43322, Waukegan, Illinois
  - Site Reference ID/Investigator# 42707, San Antonio, Texas

REFERENCES:
- [Derived] Krishnan P, Beyer J, Mistry N, Koev G, Reisch T, DeGoey D, Kati W, Campbell A, Williams L, Xie W, Setze C, Molla A, Collins C, Pilot-Matias T. In vitro and in vivo antiviral activity and resistance profile of ombitasvir, an inhibitor of hepatitis C virus NS5A. Antimicrob Agents Chemother. 2015 Feb;59(2):979-87. doi: 10.1128/AAC.04226-14. Epub 2014 Dec 1. PMID 25451055